CLINICAL TRIAL: NCT01402414
Title: Study Comparing the Effectiveness of Narrow-band UVB vs. Bath-PUVA and Narrow-band UVB + Salt Water Baths in Atopic Dermatitis
Brief Title: Narrow-band (NB)-UVB vs. Bath-PUVA and NB-UVB Plus Salt Water Baths in Atopic Dermatitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties with the Recruitement
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Sarah Terras, Thilo Gambichler, Professor, Ruhr University Bochum, Ruhr University of Bochum
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RUB-126
Record Dates: First submitted 2011-07-19; First posted 2011-07-26 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; NB-UVB; phototherapy; balneophototherapy; Bath-PUVA; SCORAD index
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NB-UVB (Active Comparator): NB-UVB irradiations adapted to the NB-MED-UVB (70%) started and increased by 10-20% per session.
  Interventions: Radiation: NB-UVB
- Bath-PUVA (Active Comparator): Phototherapy with UVA irradiation following bathing in psoralen water
  Interventions: Radiation: Bath-PUVA
- NB-UVB plus salt water baths (Active Comparator): Balneophototherapy with NB-UVB and 3% Dead Sea salt water baths
  Interventions: Radiation: NB-UVB plus salt water baths

INTERVENTIONS:
Radiation: NB-UVB — The SB-UVB irradiations (Cosmedico, Villingen-Schwenningen) are adapted to the SB-MED-UVB (70%) started and increased by 10-20% per session. The UV irradiations are carried out four times a week over a period of 4 weeks.
  Arms: NB-UVB
Radiation: Bath-PUVA — Bath PUVA is performed with 8-Methoxypsoralen baths (concentration of ultimately 0.5 mg / l ) at 37 ° C with a bath time of 20 minutes and subsequent UVA irradiation (Waldmann cabine, 320-400 nm). The first dose is 70% of MPD, followed by 20% increase. The latter takes place at the earliest after 72 hours. The UV irradiations are carried out four times a week over a period of 4 weeks.
  Arms: Bath-PUVA
Radiation: NB-UVB plus salt water baths — First, a 20-minute bath in 3% salt water (Dead Sea salt, 37 ° C) is taken. Thereafter, a NB-UVB irradiation is performed. The UV radiation can be administered according to established protocols. The NB-UVB irradiations (Cosmedico, Villingen-Schwenningen) are adapted to the NB-MED-UVB (70%) started and increased by 10-20% per session. The UV irradiations are carried out four times a week over a period of 4 weeks.
  Arms: NB-UVB plus salt water baths

SUMMARY:
In this controlled crossover study we aim to compare the efficacy of narrow-band UVB (NB-UVB) with bath-PUVA and NB-UVB plus salt water baths in atopic dermatitis.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a very common skin disorder that is characterized by pruritic inflammatory skin lesions, with patients usually having an individual or family history of atopic diseases in their background (e.g., allergic asthma and rhinitis). Defective skin barrier, immunological dysfunctions (type I and IV allergy), genetic disorders, and psychological factors contribute to the pathogenesis of AD. However, among these factors, CD4+ Th cells are reported to play a particularly crucial role in the pathogenesis of AD. Phototherapy is among the first-line approaches in the management of AD. In this context, a variety of studies have shown a beneficial effect of natural or artificial UV radiation in AD. Different broadband (BB) UV spectra (BB-UVA, BB-UVB, BB-UVA/BB-UVB) and combined treatment modalities such as balneophototherapy and PUVA have previously been proven to be effective in AD. A small controlled study has previously demonstrated that the combination of UVB/UVA and saltwater baths is superior to phototherapy alone. Previous data from uncontrolled studies also speak for the effectiveness of systemic psoralen plus UVA (PUVA) therapy. A controlled crossover study has shown that systemic PUVA therapy is clearly superior to UVA1 phototherapy both in terms of clinical score (SCORAD) and reduction of response time. Systemic PUVA has in relation to bath PUVA significantly greater adverse effects (eg, nausea, liver enzyme elevation, photocarcinogenesis). A direct comparison between NB-UVB and bath PUVA has only been studied by a half-side comparison in a small number of patients. Both therapies were proved equally effective. In a recent study, it has been shown a clear advantage of NB-UVB plus salt water baths in comparison to NB-UVB alone. Tolerability was comparable; both treatments showed to be safe.

A randomized observer-blinded controlled crossover trial is conducted in which patients with AD receive a 4-week course of both NB-UVB and bath-PUVA or NB-UVB plus salt water baths. Clinical efficacy is assessed using the Six Area, Six Sign, Atopic Dermatitis (SASSAD) score and a visual analogue scale for pruritus. Assessment of health-related quality of life was performed using the Skindex-29. Moreover, immunohistochemical, RT-PCR and serological studies are planned.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe disease AD with SASSAD-Score > 25
* Age > 18 years
* No topical steroids or topical/systemic antibiotics within the last 2 weeks, no systemic glucocorticosteroids or other immunosuppressive agents within the last 8 weeks, no phototherapy within the last 12 weeks before inclusion

Exclusion Criteria:

* Pregnancy or lactation
* Skin cancer or dysplastic naevi, photosensitive skin diseases, autoimmune diseases or relevant cardiovascular diseases
* Photo-skin type I according to Fitzpatrick
* severe cardiovascular disease
* intense UV radiation (tanning beds, sun exposure, phototherapy, etc.) 8 weeks before the start of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Clinical improvement after treatments using a validated SASSAD index | Evaluation at baseline and after 4-week treatment, 3 months follow-up
  Clinical improvement after treatments using a validated SASSAD index

SECONDARY OUTCOMES:
Evaluation of pruritus and sleeplessness visual analogue scales | Evaluation at baseline and after 4-week treatment, 3 months follow-up
  Evaluation of pruritus and sleeplessness using visual analogue scales with 0 being no complaints and 10 being the worst complaints imaginable
Measuring quality of life using the Skindex-29 | Evaluation at baseline and after 4-week treatment, 3 months follow-up
  Measuring patient's satisfaction / safety and quality of life using a qualified questionnaire: the Skindex-29.
Immunohistochemical, RT-PCR and serological parameters | Evaluation at baseline and after 4-week treatment
  Measuring several immunohistochemical, RT-PCR and serological parameters in skin and blood, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Thilo Gambichler, adjunct professor, Principal Investigator — Ruhr University Bochum
Locations (1):
- Department of Dermatology, Ruhr University Bochum, Bochum, North Rhine-Westphalia, Germany